CLINICAL TRIAL: NCT01419119
Title: A Study, Four Parallel Arms, Included Two Arms Open Randomisation to Different Doses of Vitamin D, for Assessment of Efficacy of Treatment With Vitamin D at Vitamin D Deficiency, Vitamin D Insufficiency and Suboptimal Levels of Vitamin D
Brief Title: Vitamin Deficiency in Immigrants, a Treatment Study
Acronym: VIDI2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Margareta Norberg, M.D. Ph.D., Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIDI 2
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-02

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D insufficiency; Cholecalciferol; D3; Parathyroid Hormone; 25-hydroxyvitamin D3; RDA, recommended daily intake (nutrition policy); Vitamin D; Hypovitaminosis-D; Pharmacologic treatment
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): Vitamin D3, 10 000 IU daily. Treatment to patients with Serum-vitamin D levels below 25 nmol/L
  Interventions: Drug: Cholecalciferol high dose at Vitamin D deficiency
- Group 2a (Experimental): Vitamin D3 2000 IU daily, one of two arms that patients with Serum-vitamin D levels between 25 nmol/L and 49 nmol/l will be randomised to
  Interventions: Drug: Cholecalciferol median dose at Vitamin D insufficiency
- Group 2b (Experimental): Vitamin D3 2000 IU weekly, one of two arms that patients with Serum-vitamin D levels between 25 nmol/L and 49 mol/l will be randomised to
  Interventions: Drug: Cholecalciferol low dose at Vitamin D deficiency
- Group 3 (Experimental): Vitamin D3, 2000 IU daily i.e. 3 drops orally once daily for 12 weeks, treatment to patients with Serum-vitamin D levels between 50 and 74 nmol/L
  Interventions: Drug: Cholecalciferol median dose at sufficient Vitamin D level

INTERVENTIONS:
Drug: Cholecalciferol high dose at Vitamin D deficiency — 10 000 IU daily i.e. 15 drops orally once daily for 12 weeks
  Other Names: Vigantol Oil 20 000 IU/ml, drops for oral use, solution
  Arms: Group 1
Drug: Cholecalciferol median dose at Vitamin D insufficiency — 2000 IU daily i.e. 3 drops orally once a day for 12 weeks,
  Other Names: Vigantol Oil 20 000 IU/ml, drops for oral use, solution
  Arms: Group 2a
Drug: Cholecalciferol low dose at Vitamin D deficiency — 2000 IU once a week i.e. 3 drops orally once a week (the same day every week) for 12 weeks,
  Other Names: Vigantol Oil 20 000 IU/ml, drops for oral use, solution
  Arms: Group 2b
Drug: Cholecalciferol median dose at sufficient Vitamin D level — 2000 IU daily i.e. 3 drops orally once daily for 12 weeks
  Other Names: Vigantol Oil 20 000 IU/ml, drops for oral use, solution
  Arms: Group 3

SUMMARY:
The purpose of this study is to determine the efficacy of different doses of vitamin D in persons, immigrated to Sweden from Middle East or Africa, with decreased S vitamin D.

DETAILED DESCRIPTION:
The participants in the study have taken part in a previous screening study. They are now asked to participate in this treatment study. At a screening visit blood samples for vitamin D3 and PTH are collected. Data regarding previous fractures, life style, exposure for sun, clothes, diet, smoking and physical activities are collected. The Vitamin D value predict the treatment dose.

ELIGIBILITY:
Inclusion Criteria:

* Serum- vitamin D below 75 nmol/L
* Men and female
* 25-65 years of age
* Born in Middle East or Africa, living in Umeå district

Exclusion Criteria:

* Hypersensitive to Cholecalciferol, cocos oil, palm kernel or rubber
* Serum D3 equal to or above75 nmol/L
* Hypercalcemia
* Renal insufficiency
* History of Kidney Calculi
* Nephrocalcinosis
* History of sarcoidosis and other Granulomatous Diseases
* Known malignancy
* Ongoing treatment with phenytoin, barbiturates, rifampicin, isoniazid
* Ongoing treatment with cardiac glycosides
* Ongoing treatment with thiazides
* Ongoing treatment with Etalpha, Rocaltrol, ergocalciferol, Dygratal
* Ongoing treatment with drugs involving fat absorption; Orlistat Colestyramin
* Oral treatment with glucocorticoids
* Ongoing treatment with Aluminum Compounds drugs
* Ongoing treatment with Omega -3, vitamin D and/or calcium
* Immobilisation
* Other medial reason not to participate according to the investigator
* Pregnancy (women with S-D3 below 25 nmol/)
* Breastfeeding

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margareta Norberg, M.D. Ph.D, Principal Investigator — Dept of Epidemiology and Global Health, Umeå University
Locations (1):
- Ålidhems hälsocentral, Umeå, Umeå, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Vitamin D3, 10 000 IU daily. Treatment to patients with Serum-vitamin D levels below 25 nmol/L
  Cholecalciferol: 10 000 IU daily i.e. 15 drops orally once daily for 12 weeks
- Group 2a: Vitamin D3 2000 IU daily, one of two arms that patients with Serum-vitamin D levels between 25 nmol/L and 49 nmol/l will be randomised to
  Cholecalciferol: 2000 IU daily i.e. 3 drops orally once a day for 12 weeks,
- Group 2b: Vitamin D3 2000 IU weekly, one of two arms that patients with Serum-vitamin D levels between 25 nmol/L and 49 mol/l will be randomised to
  Cholecalciferol: 2000 IU once a week i.e. 3 drops orally once a week (the same day every week) for 12 weeks,
- Group 3: Vitamin D3, 2000 IU daily i.e. 3 drops orally once daily for 12 weeks, treatment to patients with Serum-vitamin D levels between 50 and 74 nmol/L
  Cholecalciferol: 2000 IU daily i.e. 3 drops orally once daily for 12 weeks
Period: Overall Study
Arm/Group | Group 1 | Group 2a | Group 2b | Group 3
Started | 23 | 56 | 50 | 31
Completed | 16 | 54 | 49 | 28
Not Completed | 7 | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Only participants who completed the study protocol, i.e.analyses per protocol
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2a | Group 2b | Group 3 | Total
Number analyzed (Participants) | 16 | 54 | 49 | 28 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (11.2) | 41.3 (11.5) | 40.9 (9.8) | 43.2 (11.2) | 41.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 26 | 23 | 14 | 68
  Male | 11 | 28 | 26 | 14 | 79
Region of Enrollment [Number; unit: participants]
  Sweden | 16 | 54 | 49 | 28 | 147

OUTCOME MEASURES:

1. Primary Outcome: Serum-vitamin D
Description: Levels of serum vitamin D3
Time Frame: Baseline
Population: Participants who completed the study protocol
Measure: Mean (Standard Deviation); unit: 25(OH)D, nmol/L
Arm/Group | Group 1 | Group 2a | Group 2b | Group 3
Number analyzed (Participants) | 16 | 54 | 49 | 28
25(OH)D, nmol/L | 19.7 (4.0) | 34.4 (6.5) | 38.7 (6.5) | 58.7 (6.3)
Statistical Analysis 1: Comparison: Group 1 vs Group 2a vs Group 2b vs Group 3; Test type: Superiority; p = 0.001, t-test, 2 sided

2. Primary Outcome: Level of Vitamin D at End of the Treatment Period of 12 Weeks
Description: Serum Vitamin D, 25-(OH)D
Time Frame: End of treatment period 12 weeks after baseline
Measure: Mean (Standard Deviation); unit: 25(OH)D, nmol/L
Arm/Group | Group 1 | Group 2a | Group 2b | Group 3
Number analyzed (Participants) | 16 | 54 | 49 | 28
25(OH)D, nmol/L | 140.8 (31.9) | 72.5 (14.6) | 52.3 (9.9) | 81.0 (14.8)
Statistical Analysis 1: Comparison: Group 1 vs Group 2a vs Group 2b vs Group 3; Test type: Superiority; p = 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: The treatment period of 12 weeks
Arm/Group | Group 1 | Group 2a | Group 2b | Group 3
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/56 | 0/50 | 0/31
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/56 | 0/50 | 0/31
Other Adverse Events (participants affected / at risk) | 8/23 | 19/56 | 12/50 | 5/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=23) | Group 2a (N=56) | Group 2b (N=50) | Group 3 (N=31)
Suspected serious adverse event (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Mental agitation. The subject doubled the study medication concomitantly with changes of anti-depressant medication. Unclear whether symptoms wer due to a rapid increase to high serum 25(OH)D levels or the anti-depressive medication.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=23) | Group 2a (N=56) | Group 2b (N=50) | Group 3 (N=31)
Adverse Events (General disorders) | 8 (8) | 19 (19) | 12 (12) | 5 (5) — The AEs were miscellaneous and mild without any clear pattern, while four were due to other causes or conditions that were known before the study. Examples: obstipation, headache, pain in the wrists

LIMITATIONS AND CAVEATS:
This open partly RCT was conducted during September 2011-May 2012 at the Umeå University Hospital Clinical Research Centre, monitored by the Clinical Trial Unit, Region Västerbotten, Sweden. The study treatment was vitamin D supplementation (25(OH)D) during 12 weeks.

The trial was reported to the Swedish Medical Products Agency in August 2013 and to the European Medicines Agency in November 2021. No reports have been accepted to publication in Scientific journals

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes